CLINICAL TRIAL: NCT05032898
Title: Acute Exacerbation of Chronic Obstructive Pulmonary Disease Inpatient Registry Study Stage II
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Chen Wang, Principal investigator, China-Japan Friendship Hospital
Other Study IDs: AECOPD-IRS-II
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: registries; demography; therapeutics; disease management; mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to provide high quality data and give a comprehensive overview of characteristics, clinical features, management and prognosis during exacerbations and stable periods among inpatients with acute exacerbation of chronic obstructive pulmonary disease in real-world China.

DETAILED DESCRIPTION:
Objective: The aim of this study is to provide high quality data and give a comprehensive overview of characteristics, clinical features, management and prognosis during exacerbations and stable periods among inpatients with acute exacerbation of chronic obstructive pulmonary disease in real-world China.

Eligibility Criteria: Details are shown in the Eligibility Criteria part.

Procedures and Measurements: At admission, each eligible subject will be given an in-depth interview to collect the demographics, smoking history, medical history, management of disease during stable period, etc. During hospitalization, treatment and auxiliary examination results including laboratory and lung function tests will be recorded if available. To ensure the quality and uniformity of spirometry data, training on performing spirometry will be provided to each study site by professional doctors from central site. At discharge, physicians will record the discharge diagnoses and clinical outcomes including death, intensive care unit admission, chronic obstructive pulmonary disease assessment test (CAT) score and total direct cost for each participant. During follow-ups, clinical outcomes including death and exacerbation events, change of medication, new-developed complications, auxiliary examination results, and economic burden will be collected.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* hospitalized with main diagnosis of acute exacerbation of chronic obstructive pulmonary disease (AECOPD)

Exclusion Criteria:

* refusing to sign informed consent forms
* participating in clinical trials or intervention studies of drugs
* diagnosed as active pulmonary tuberculosis, or acute left heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with acute exacerbation of chronic obstructive pulmonary disease will be consecutively recruited from target hospitals.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
All-cause in-hospital mortality | From date of admission to date of discharge, an expected median of 10 days
  All-cause mortality during hospitalization
Incidence of readmission due to acute exacerbation of chronic obstructive pulmonary disease within 30 days after discharge | 30 days after day of discharge
  Incidence of readmission due to acute exacerbation of chronic obstructive pulmonary disease (AECOPD) within 30 days after discharge

SECONDARY OUTCOMES:
All-cause mortality | 30 days and 1 year after day of discharge
  All-cause mortality during follow-ups
Incidence of readmission due to acute exacerbation of chronic obstructive pulmonary disease within 1 year after discharge | 1 year after day of discharge
  Incidence of readmission due to acute exacerbation of chronic obstructive pulmonary disease (AECOPD) within 1 year after discharge
Time to the first readmission due to acute exacerbation of chronic obstructive pulmonary disease | 30 days, 1 year after day of discharge
  Time to the first readmission due to acute exacerbation of chronic obstructive pulmonary disease (AECOPD) during follow-ups
Post-bronchodilator forced expiratory volume in one second (L) | 30 days, 1 year after day of discharge
  Post-bronchodilator forced expiratory volume in one second (L) during follow-ups
Predicted post-bronchodilator forced expiratory volume in one second (%) | 30 days, 1 year after day of discharge
  Predicted post-bronchodilator forced expiratory volume in one second (%) during follow-ups
Post-bronchodilator forced vital capacity (L) | 30 days, 1 year after day of discharge
  Post-bronchodilator forced vital capacity (L) during follow-ups
Post-bronchodilator forced expiratory volume in one second to forced vital capacity | 30 days, 1 year after day of discharge
  Post-bronchodilator forced expiratory volume in one second to forced vital capacity during follow-ups
Chronic obstructive pulmonary disease assessment test (CAT) score | At day of discharge (an expected median of 10 days), 30 days, 1 year after day of discharge
  Chronic obstructive pulmonary disease assessment test (CAT) score at day of discharge and during follow-ups. CAT is an 8-item questionnaire used to measure the impact of respiratory disease on patients' health status. The score of CAT ranges from 0 to 40, with 0 indicating the best health status while 40 as the worst.
Modified medical research council (mMRC) dyspnea scale | At day of discharge (an expected median of 10 days), 30 days, 1 year after day of discharge
  Modified medical research council (mMRC) dyspnea scale at day of discharge and during follow-ups. mMRC includes 5 grades (0, 1, 2, 3 and 4), where higher grade reflects worse health-related quality of life and higher symptom burden.
Direct total cost of chronic obstructive pulmonary disease management | At day of discharge (an expected median of 10 days), 30 days, 1 year after day of discharge
  Direct total cost of chronic obstructive pulmonary disease management during hospitalization and follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Doctor, Study Chair — Institue of Basic Medical Sciences Chinese Academy of Medical Sciences; Ting Yang, Doctor, Principal Investigator — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results (text, tables, figures, and appendices) reported in the publication of summary data, study protocol, statistical analysis plan (SAP), analytic code will be shared from 1 to 3 years following the completion of data cleaning. All above could be shared with researches who provide a methodologically sound and feasible proposal approved by principal investigator (email address: cyh-birm@263.net, dryangting@qq.com) and a signed data access agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: From 1 to 3 years following the completion of data cleaning.
Access Criteria: Researches should send a proposal to cyh-birm@263.net or dryangting@qq.com. If the proposal is methodologically sound, feasible and approved by the principal investigator, data requestor could gain access after signing a data access agreement.